CLINICAL TRIAL: NCT00666224
Title: A Multinational, Multicenter, Randomized, Double-Blind, Placebo Controlled, Parallel Group Study to Evaluate the Effect of Early Glatiramer Acetate Treatment in Delaying the Conversion to Clinically Definite Multiple Sclerosis (CDMS) of Subjects Presenting With Clinically Isolated Syndrome (CIS)
Brief Title: Evaluate Early Glatiramer Acetate Treatment in Delaying Conversion to Clinically Definite Multiple Sclerosis of Subjects Presenting With Clinically Isolated Syndrome
Acronym: PreCISe
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GA 9010
Record Dates: First submitted 2008-04-22; First posted 2008-04-24 (Estimated); Results first posted 2012-06-13 (Estimated); Last update posted 2012-06-25 (Estimated); Status verified 2012-06

CONDITIONS: Multiple Sclerosis
Keywords: Clinically Definite Multiple Sclerosis; Clinically Isolated Syndrome; Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Glatiramer Acetate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Glatiramer acetate (Experimental): Glatiramer acetate 20 mg once daily by subcutaneous injection is administered in both the double-blind and open label periods.
  Interventions: Drug: Glatiramer Acetate (DB); Drug: Glatiramer Acetate (OL)
- Placebo (DB) to GA (OL) (Placebo Comparator): Placebo matching glatiramer acetate once daily by subcutaneous injection during the double-blind period (DB). Glatiramer acetate (GA) 20 mg once daily by subcutaneous injection during the open-label period (OL).
  Interventions: Drug: Placebo; Drug: Glatiramer Acetate (OL)

INTERVENTIONS:
Drug: Glatiramer Acetate (DB) — Double blind period (DB): glatiramer acetate (GA) by subcutaneous injection, 20mg, once daily, for up to 36 months or until conversion to clinically definite multiple sclerosis (CDMS).
  Other Names: Copaxone®
  Arms: Glatiramer acetate
Drug: Placebo — Double blind period (DB): subcutaneous injection of placebo, once daily, for up to 36 months or until conversion to CDMS
  Arms: Placebo (DB) to GA (OL)
Drug: Glatiramer Acetate (OL) — Open label period (OL): glatiramer acetate (GA), 20 mg, subcutaneous injection, once daily, given for up to an additional 24 months.
  Other Names: Copaxone®

SUMMARY:
The primary objective is to assess the effect of treatment with glatiramer acetate (GA) compared to placebo on the time to conversion to CDMS, as determined by Poser criteria (the occurrence of the second clinical attack) during the double-blind period. The secondary objective is to assess, within the time frame of the up to 3-year double-blind, placebo-controlled study period, the effect of GA on clinical and Magnetic Resonance Imaging (MRI) parameters. The long-term objectives of the study (exploratory in nature) are to assess, within the time frame of 5 years, the neuroprotective effect of early versus delayed treatment with GA as reflected by clinical and MRI parameters measuring the accumulated irreversible brain tissue damage.

A pre-planned interim analysis was performed on all efficacy and safety data accumulated in the database up to October 14, 2007, i.e. when 81% of exposure to treatment in the double-blind, placebo-controlled period had been collected. Upon review of the interim analysis results, the Data Monitoring Committee (DMC) recommended that the double-blind portion of the study be stopped and that subjects be switched to the 2-year Open-label period, during which time they would have the option of receiving GA therapy. The sponsor (Teva) adopted the DMC recommendations and took the necessary action towards its implementation.

ELIGIBILITY:
Inclusion Criteria:

1. The subject must have undergone a single clinical attack.
2. The subject must have a unifocal clinical presentation.
3. The subject should be enrolled within the period of 90 days after onset of a single unifocal clinical attack (index attack).
4. There must be 2 or more cerebral lesions highly suspicious of multiple sclerosis (MS) on the screening Magnetic Resonance Imaging (MRI), measuring 6mm or more in diameter.
5. Subjects must be between the ages of 18 and 45 years inclusive.
6. Subjects must not have taken corticosteroids within the 30 days prior to the MRI at the baseline visit.
7. Subjects may be male or female. Women of child-bearing potential must practice a medically acceptable method of birth control. Acceptable methods include oral contraceptive, contraceptive patch, long-acting injectable contraceptive, or double-barrier method (condom or intrauterine device with spermicide).
8. The subjects must be willing and able to give written informed consent, prior to entering the study.

Exclusion Criteria:

1. Multifocal clinical presentation.
2. Diseases other than MS responsible for the clinical/MRI presentation. The following laboratory tests must be part of the subject's medical history for differential diagnosis of clinically isolated syndrome (CIS): erythrocyte sedimentation rate (ESR), antinuclear antibody (ANA), complement (C3, C4) and anticardiolipin IgG - IgM. In the event that the results of these tests are inconclusive, the following additional tests may be requested by the Eligibility Evaluation Committee: syphilis screening, vitamin B12 and folic acid. In the case of spinal cord CIS presentation, a spinal cord MRI is required for confirmation of diagnosis in the medical history of the subject.
3. Use of experimental or investigational drugs, including IV immunoglobulin, and/or participation in an investigational drug study within 6 months prior to study entry.
4. Use of interferon agents within 6 months prior to the screening visit.
5. Chronic corticosteroid treatment (more than 30 consecutive days) in the 6 months prior to study entry.
6. Pregnancy or breast feeding.
7. Subjects who experience a relapse between the screening (month -1) and baseline (month 0) visits.
8. Life-threatening or other clinically significant disease.
9. A medical or psychiatric condition that affects the subject's ability to give informed consent, or to complete the study, or if the subject is considered by the treating neurologist/physician to be, for any other reason, an unsuitable candidate for this study.
10. A known history of sensitivity to mannitol.
11. A known history of sensitivity to gadolinium.
12. Inability to successfully undergo MRI scanning.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 481 (Actual)
Dates: Start 2004-01; Primary Completion 2007-10 (Actual); Study Completion 2010-06 (Actual)

REFERENCES:
- [Result] Comi G, Martinelli V, Rodegher M, Moiola L, Bajenaru O, Carra A, Elovaara I, Fazekas F, Hartung HP, Hillert J, King J, Komoly S, Lubetzki C, Montalban X, Myhr KM, Ravnborg M, Rieckmann P, Wynn D, Young C, Filippi M; PreCISe study group. Effect of glatiramer acetate on conversion to clinically definite multiple sclerosis in patients with clinically isolated syndrome (PreCISe study): a randomised, double-blind, placebo-controlled trial. Lancet. 2009 Oct 31;374(9700):1503-11. doi: 10.1016/S0140-6736(09)61259-9. Epub 2009 Oct 6. PMID 19815268

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A clinically isolated syndrome (CIS) is a first neurological episode, lasting at least 24 hours, caused by inflammation/demyelination in one or more sites in the central nervous system (CNS.) Subjects were enrolled within 90 days of the event and randomized up to 32 days following screening.
Pre-assignment Details: Six-hundred and nineteen (619) subjects were screened for this study; 138 subjects were screening failures, including one subject, randomized in error. This subject, who had a relapse between screening visit and baseline, never received any treatment, and is considered a screening failure.
Groups:
- Glatiramer Acetate: Glatiramer acetate (GA) 20 mg once daily by subcutaneous injection during the double-blind period. Following a pre-planned interim analysis, the Data Monitoring Committee (DMC) recommended that the double blind period be closed and participants moved into the Open Label (OL) period. Participants in this treatment arm continued taking glatiramer acetate 20 mg once daily by subcutaneous injection during the open-label (OL) period.
- Placebo (DB) to GA (OL): Placebo matching glatiramer acetate given once daily by subcutaneous injection during the double-blind period (DB). Following a pre-planned interim analysis, the Data Monitoring Committee (DMC) recommended that the double blind period be closed and participants moved into the Open Label (OL) period. Glatiramer acetate (GA) given 20 mg once daily by subcutaneous injection during the open-label period (OL).
Period: Double-Blind
Arm/Group | Glatiramer Acetate | Placebo (DB) to GA (OL)
Started | 243 | 238
Completed | 198 (78 completed 3 years treatment, 66 converted to CDMS, 54 switched to OL as per DMC) | 211 (55 completed 3 years treatment, 109 converted to CDMS, 47 switched to OL as per DMC)
Not Completed | 45 | 27
Not completed — Adverse Event | 15 | 5
Not completed — Lost to Follow-up | 2 | 2
Not completed — Withdrawal by Subject | 18 | 14
Not completed — Physician Decision | 0 | 3
Not completed — Sponsor decision | 1 | 0
Not completed — Pregnancy | 3 | 2
Not completed — Noncompliance | 1 | 0
Not completed — Death | 1 | 0
Not completed — Undefined/Unknown | 4 | 1
Period: Open-Label
Arm/Group | Glatiramer Acetate | Placebo (DB) to GA (OL)
Started | 198 (454 participants took at least one dose of GA including 45 who didn't continue into the OL.) | 211
Completed | 163 | 126
Not Completed | 35 | 85
Not completed — Adverse Event | 8 | 43
Not completed — Lost to Follow-up | 4 | 5
Not completed — Withdrawal by Subject | 12 | 25
Not completed — Physician Decision | 7 | 5
Not completed — Pregnancy | 1 | 5
Not completed — Noncompliance | 2 | 1
Not completed — Undefined/Unknown | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Glatiramer Acetate (Double-blind Period): Glatiramer acetate 20 mg once daily by subcutaneous injection during the double-blind period.
- Placebo (Double-blind Period): Placebo matching GA once daily by subcutaneous injection during the double-blind period.
- Total: Total of all reporting groups
Arm/Group | Glatiramer Acetate (Double-blind Period) | Placebo (Double-blind Period) | Total
Number analyzed (Participants) | 243 | 238 | 481
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 243 | 238 | 481
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 31.5 (6.9) | 30.8 (7.0) | 31.2 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 159 | 163 | 322
  Male | 84 | 75 | 159
Race/Ethnicity, Customized [Number; unit: participants]
  Asian / Oriental | 2 | 1 | 3
  Black or African American | 1 | 1 | 2
  Caucasian | 233 | 229 | 462
  Hispanic | 3 | 2 | 5
  Other (not specified) | 4 | 5 | 9
Region of Enrollment [Number; unit: participants]
  Argentina | 7 | 6 | 13
  Australia | 7 | 6 | 13
  Austria | 5 | 6 | 11
  Denmark | 5 | 6 | 11
  Finland | 10 | 10 | 20
  France | 11 | 11 | 22
  Germany | 32 | 31 | 63
  Hungary | 16 | 15 | 31
  Italy | 56 | 57 | 113
  New Zealand | 4 | 3 | 7
  Norway | 2 | 2 | 4
  Romania | 28 | 30 | 58
  Spain | 23 | 22 | 45
  Sweden | 2 | 0 | 2
  United Kingdom | 15 | 12 | 27
  United States | 20 | 21 | 41
Participants Who Used Corticosteroids for Initial Attack [Number; unit: participants]
  Used corticosteroids | 149 | 159 | 308
  Did not use corticosteroids | 94 | 79 | 173

OUTCOME MEASURES:

1. Primary Outcome: Time to Clinically Definite Multiple Sclerosis (CDMS) Conversion
Description: Data from interim analysis with database lock on October 14, 2007. The time from randomization to conversion to CDMS as determined by the occurrence of a second clinical attack during the double-blind period. Poser criteria are: Two relapses and clinical evidence of two separate lesions; clinical evidence of one lesion and paraclinical evidence of another separate lesion. The two relapses must involve different parts of Central Nervous System and must be separated by a period of at least one month. Lesions are determined by Magnetic Resonance Imaging (MRI).
Time Frame: up to 3 years
Population: Intent-to-Treat (ITT) analysis set. The ITT consists of all participants who have been randomized and received at least one dose of glatiramer acetate or placebo.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Glatiramer Acetate (Double-blind Period) | Placebo (Double-blind Period)
Number analyzed (Participants) | 243 | 238
days | 657.85 (349.3) | 590.54 (340.2)
Statistical Analysis 1: Comparison: Glatiramer Acetate (Double-blind Period) vs Placebo (Double-blind Period); Test type: Superiority or Other; p = 0.0005, Regression, Cox — Type of unifocal presentation at baseline, past corticosteroid treatment (Yes/No) for the initial attack prior to randomization, and center effects as covariates; Cox Proportional Hazard = 0.55, 95% CI 2-sided [0.40 to 0.77]

2. Secondary Outcome: Number of New T2 Brain Lesions Observed at the Last Observed Value (LOV) in the Double-blind Period
Description: Data from interim analysis with database lock on October 14, 2007. T2 lesions are brain lesions that show on magnetic resonance imaging (MRI) and are associated with multiple sclerosis. This outcome measures the number of new lesions at the last observed value. Last Observed Value (LOV) is defined as the last post baseline measurement taken on study drug but no more than 30 days after study drug cessation.
Time Frame: up to 3 years
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: new T2 lesions
Arm/Group | Glatiramer Acetate (Double-blind Period) | Placebo (Double-blind Period)
Number analyzed (Participants) | 243 | 238
new T2 lesions | 0.7 (1.7) | 1.8 (3.6)
Statistical Analysis 1: Comparison: Glatiramer Acetate (Double-blind Period) vs Placebo (Double-blind Period); Test type: Superiority or Other; p < 0.0001, Quasi-Likelihood NB* Regression; *NB = Negative Binomial Center and baseline number of enhancing lesions as covariates; Rate ratio = 0.42, 95% CI 2-sided [0.29 to 0.61]

3. Secondary Outcome: Change From Baseline to Last Observed Value (LOV) in T2 Brain Lesion Volume in the Double-blind Period
Description: Data from interim analysis with database lock on October 14, 2007. The difference in T2 brain lesion volume as observed in MRIs from baseline to the last observed value. Last Observed Value (LOV) is defined as the last post baseline measurement taken on study drug but no more than 30 days after study drug cessation.
Time Frame: Day 0 (baseline), up to 3 years
Population: Intent to treat population for which data at both timepoints are available
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Glatiramer Acetate (Double-blind Period) | Placebo (Double-blind Period)
Number analyzed (Participants) | 218 | 221
ml | 1.2 (2.6) | 2.6 (3.9)
Statistical Analysis 1: Comparison: Glatiramer Acetate (Double-blind Period) vs Placebo (Double-blind Period); Test type: Superiority or Other; p = 0.0013, ANCOVA; Used log-transformed measurements comparing the adjusted geometric means of T2 volume. Center and baseline T2 volume used as covariates; Geometric means ratio = 0.87, 95% CI 2-sided [0.79 to 0.95]

4. Secondary Outcome: Percentage Change in Brain Volume From Baseline to the Last Observed Value (LOV) During the Double-blind Period Using the Structural Image Evaluation of Normalized Atrophy (SIENA) Technique
Description: Data from interim analysis with database lock on October 14, 2007. Brain volume was measured annually by magnetic resonance imaging (MRI) during the Double-blind period. Brain atrophy was measured by comparing the change in brain volume from baseline to the Last Observed Value (LOV). LOV is defined as the last post baseline measurement taken on study drug but no more than 30 days after study drug cessation. SIENA is a fully automated method of analyzing longitudinal brain change.
Time Frame: Day 0 (baseline), up to 3 years
Population: Intent to treat population of participants with both baseline and last observed values.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Glatiramer Acetate (Double-blind Period) | Placebo (Double-blind Period)
Number analyzed (Participants) | 191 | 174
percent change | -0.3 (0.6) | -0.4 (0.7)

5. Primary Outcome: Twenty-fifth Percentile (25%) Kaplan-Meier Estimates for Time From Randomization to Conversion to Clinically Definite Multiple Sclerosis (CDMS) During the Double-blind Period
Description: Data from interim analysis with database lock on October 14, 2007. Due to the number of participants in the glatiramer acetate group that converted to CDMS (see outcome #6), the 25th percentile was considered when running the Kaplan-Meier estimate for time to conversion to CDMS. Conversion to CDMS is determined by the occurrence of the second clinical attack.
Time Frame: up to 3 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: days
Arm/Group | Glatiramer Acetate (Double-blind Period) | Placebo (Double-blind Period)
Number analyzed (Participants) | 243 | 238
days | 722 [505 to NA] — Not able to be estimated due to small numbers of participants converting to CDMS | 336 [260 to 456]

6. Secondary Outcome: Percentage of Participants Who Converted to Clinically Definite Multiple Sclerosis (CDMS) During the Double-blind Period
Description: Data from interim analysis with database lock on October 14, 2007. Conversion to CDMS as determined by the occurrence of a second clinical attack during the double-blind period. Poser criteria are: Two relapses and clinical evidence of two separate lesions; clinical evidence of one lesion and paraclinical evidence of another separate lesion. The two relapses must involve different parts of Central Nervous System and must be separated by a period of at least one month. Lesions are determined by Magnetic Resonance Imaging (MRI).
Time Frame: up to 3 years
Population: Intent-to-Treat (ITT) analysis set.
Measure: Number; unit: percentage of total participants
Arm/Group | Glatiramer Acetate (Double-blind Period) | Placebo (Double-blind Period)
Number analyzed (Participants) | 243 | 238
percentage of total participants | 24.7 | 42.9
Statistical Analysis 1: Comparison: Glatiramer Acetate (Double-blind Period) vs Placebo (Double-blind Period); Test type: Superiority or Other; p < 0.0001, Regression, Logistic — Type of unifocal presentation, past corticosteroid treatment (Yes/No) for the initial attack prior to randomization and center effects as covariates; Odds Ratio (OR) = 0.41, 95% CI 2-sided [0.27 to 0.61]

ADVERSE EVENTS:
Time Frame: The double-blind period was up to three years. The entire study included the double-blind period (up to three years) and the open-label period (up to an additional two years).
Groups:
- Glatiramer Acetate (Double-blind Period): Glatiramer acetate 20 mg once daily by subcutaneous injection during the double-blind period. This subset of the GA treatment experience allows for comparison to the Placebo Double-blind Period data.
- Glatiramer Acetate (Entire Study): Glatiramer acetate (GA) 20 mg once daily by subcutaneous injection. GA adverse experiences from both the double-blind and open-label periods are combined in this column.
Arm/Group | Placebo (Double-blind Period) | Glatiramer Acetate (Double-blind Period) | Glatiramer Acetate (Entire Study)
Serious Adverse Events (participants affected / at risk) | 19/238 | 11/243 | 44/454
Other Adverse Events (participants affected / at risk) | 165/238 | 191/243 | 352/454
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Double-blind Period) (N=238) | Glatiramer Acetate (Double-blind Period) (N=243) | Glatiramer Acetate (Entire Study) (N=454)
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 1
Hydrocele (Congenital, familial and genetic disorders) | 1 | 0 | 0
Deafness (Ear and labyrinth disorders) | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal tenderness (Gastrointestinal disorders) | 0 | 1 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 2
Chills (General disorders) | 0 | 0 | 1
Feeling Hot (General disorders) | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1
Anaphylactic Reaction (Immune system disorders) | 0 | 0 | 4
Anaphylactic shock (Immune system disorders) | 0 | 0 | 1
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 1 | 2
Appendicitis (Infections and infestations) | 0 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Avulsion fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Multiple drug overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1
Renal injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 2
Platelet count decreased (Investigations) | 0 | 1 | 1
Transaminases increased (Investigations) | 1 | 0 | 0
Visual field tests abnormal (Investigations) | 0 | 1 | 1
Fistula (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Rectal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Amnesia (Nervous system disorders) | 1 | 0 | 0
Aphasia (Nervous system disorders) | 1 | 0 | 0
Cluster headache (Nervous system disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1
Facial palsy (Nervous system disorders) | 1 | 0 | 0
Intracranial venous sinus thrombosis (Nervous system disorders) | 0 | 0 | 1
Multiple sclerosis relapse (Nervous system disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 1 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1
Imminent abortion (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 1
Completed suicide (Psychiatric disorders) | 0 | 1 | 1
Depression (Psychiatric disorders) | 1 | 0 | 1
Suicide attempt (Psychiatric disorders) | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 1
Renal colic (Renal and urinary disorders) | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 2
Abortion induced (Surgical and medical procedures) | 1 | 0 | 0
Anal fissure excision (Surgical and medical procedures) | 1 | 0 | 0
Appendicectomy (Surgical and medical procedures) | 1 | 0 | 0
Bladder neoplasm surgery (Surgical and medical procedures) | 0 | 0 | 1
Breast reconstruction (Surgical and medical procedures) | 1 | 0 | 0
Cholecystectomy (Surgical and medical procedures) | 0 | 1 | 2
Cholesteatoma removal (Surgical and medical procedures) | 0 | 1 | 1
Endometrial ablation (Surgical and medical procedures) | 1 | 0 | 0
Haemorrhoid operation (Surgical and medical procedures) | 0 | 0 | 1
Lipoma excision (Surgical and medical procedures) | 0 | 0 | 1
Nail operation (Surgical and medical procedures) | 1 | 0 | 0
Resection of rectum (Surgical and medical procedures) | 0 | 0 | 1
Skin neoplasm excision (Surgical and medical procedures) | 0 | 1 | 1
Tonsillectomy (Surgical and medical procedures) | 0 | 0 | 1
Flushing (Vascular disorders) | 0 | 0 | 1
Varicose vein (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5.0% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Double-blind Period) (N=238) | Glatiramer Acetate (Double-blind Period) (N=243) | Glatiramer Acetate (Entire Study) (N=454)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 13 | 28
Tachycardia (Cardiac disorders) | 0 | 10 | 25
Diarrhoea (Gastrointestinal disorders) | 10 | 11 | 26
Nausea (Gastrointestinal disorders) | 12 | 18 | 34
Vomiting (Gastrointestinal disorders) | 5 | 15 | 29
Chest discomfort (General disorders) | 1 | 13 | 25
Fatigue (General disorders) | 22 | 26 | 40
Injection site erythema (General disorders) | 15 | 72 | 140
Injection site haematoma (General disorders) | 22 | 16 | 22
Injection site induration (General disorders) | 3 | 25 | 45
Injection site pain (General disorders) | 18 | 54 | 105
Injection site pruritus (General disorders) | 4 | 31 | 58
Injection site reaction (General disorders) | 5 | 25 | 41
Injection site swelling (General disorders) | 6 | 24 | 53
Pyrexia (General disorders) | 16 | 13 | 31
Bronchitis (Infections and infestations) | 8 | 12 | 28
Influenza (Infections and infestations) | 34 | 27 | 55
Nasopharyngitis (Infections and infestations) | 49 | 48 | 94
Pharyngitis (Infections and infestations) | 19 | 17 | 32
Rhinitis (Infections and infestations) | 8 | 14 | 23
Sinusitis (Infections and infestations) | 12 | 15 | 30
Tonsillitis (Infections and infestations) | 7 | 11 | 23
Upper respiratory tract infection (Infections and infestations) | 16 | 22 | 41
Urinary tract infection (Infections and infestations) | 11 | 10 | 33
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 9 | 29
Back pain (Musculoskeletal and connective tissue disorders) | 19 | 25 | 47
Pain in extremity (Musculoskeletal and connective tissue disorders) | 17 | 13 | 28
Headache (Nervous system disorders) | 43 | 54 | 80
Paraesthesia (Nervous system disorders) | 18 | 21 | 37
Anxiety (Psychiatric disorders) | 12 | 15 | 30
Depression (Psychiatric disorders) | 14 | 17 | 35
Cough (Respiratory, thoracic and mediastinal disorders) | 14 | 19 | 30
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 18 | 48
Erythema (Skin and subcutaneous tissue disorders) | 4 | 11 | 28
Flushing (Vascular disorders) | 1 | 15 | 31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Should the investigator wish to publish the results of this study, he/she agrees to provide Teva with a manuscript for review 60 days prior to submission for publication. Teva retains the right to delete confidential information and to object to suggest publication and/or its timing (at the Company's sole discretion).

If Teva chooses to publish this study a copy will be provided to the investigator at least 30 days prior to the expected date of submission to the intended publisher.